CLINICAL TRIAL: NCT00634972
Title: Topical Application of ACULAR a Randomized, Vehicle Controlled Clinical Trial: Efficiency in Inhibiting Proliferative Retinopathy of Prematurity
Brief Title: Efficient Study of ACULAR in Inhibiting Proliferative Retinopathy in Prematurity
Acronym: ROP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study could not be completed as the company producing this product interrupted their supply of this medication
Sponsor: University of South Alabama (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 05-156; 05-156
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Retinopathy of Prematurity; Retinal Detachment; Blindness
Keywords: Retinopathy of Prematurity; Premature Infants; ACULAR; Refresh Tears
MeSH Terms: conditions — Retinopathy of Prematurity; Retinal Detachment; Blindness; Premature Birth | interventions — Ketorolac Tromethamine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ACULAR; Drug: REFRESH TEARS
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ACULAR — infants enrolled in the study will receive 1 drop of the ROP Study drug in each eye 3 times a day (every 8 hours.
  Other Names: Acular LS 0.4% 5 mL; - from Allergan
  Arms: 1
Drug: REFRESH TEARS — infants enrolled in the study will receive 1 drop of the ROP Study drug in each eye 3 times a day (every 8 hours.
  Other Names: REFRESH TEARS 0.1 fl oz; - from Allergan
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
The purpose of this study is to test whether ACULAR, a nonsteroidal anti-inflammatory eye drop medication, can prevent the development of retinopathy of prematurity (ROP) and/ or decrease its severity.In this study ACULAR will be compared to a placebo (artificial tear).

The hypothesis would be that ACULAR treatment will decrease the incidence of moderate to severe ROP (grade II and above)by 50%.

DETAILED DESCRIPTION:
Each year ROP affects an estimated 14,000-16,000 premature, low birth weight infants in the United States and thousands more worldwide, making it a leading cause of vision loss in children. Of these cases, approximately 1500 infants will develop severe ROP that requires surgical treatment. Despite those treatment, about 400-600 infants with severe ROP still become legally blind each year.

ACULAR® (Ketorolac eye drop) is a member of nonsteroidal anti-inflammatory drugs (NSAIDs) available for toipcal ocular use. ACULAR acts as prostaglandin inhibitor and as such decrease prostaglandin E2 production. An increase in prostaglandin production has been associated with various inflammatory eye disease.For instance ACULAR has been shown to be effective in preventing the post cataract surgery inflammation that result in macular edema in adults. Activation of the prostaglandin cascade has been demonstrated in animal models of ROP. A previous non randomized study using ACULAR for ROP prevention has shown a possible beneficial effect and no observed adverse effect. To clearly demonstrated and confirm this finding a randomized study is thus necessary before one can advocate its use for prevention of ROP.The medication is FDA approved in pediatrics for allergic conjunctivitis and post surgical ocular inflammation.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants of gestational age less or equal to 28 weeks completed gestational age and 10 to 15 days of postnatal age admitted to our regional NICU

Ages: 10 Days to 15 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabien G Eyal, M.D., Principal Investigator — University Of South Alabama, Children's & Women's Hospital
Locations (1):
- Division of Neonatology, Children's & Women's Hospital, University of South Alabama, Mobile, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Drop of the ROP Study Drug: ACULAR: infants enrolled in the study will receive 1 drop of the ROP Study drug in each eye 3 times a day (every 8 hours.
  REFRESH TEARS: infants enrolled in the study will receive 1 drop of the ROP Study drug in each eye 3 times a day (every 8 hours.
- Placebo: placebo
Period: Overall Study
Arm/Group | 1 Drop of the ROP Study Drug | Placebo
Started | 40 | 43
Completed | 40 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Drop of the ROP Study Drug | Placebo | Total
Number analyzed (Participants) | 40 | 43 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 43 | 83
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 18 | 24 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of ACULAR Compared to Placebo in Inhibiting the Development of Retinopahty of Prematurity in a High Risk Very Immature Preterm Group of Infants
Time Frame: 3-4 years
Population: The study was prematurely interrupted. As we could not achieve the recruitment of a sufficient number of patients that was required to reach the preplanned power for a statistically significant results, no data analysis was completed.
Arm/Group | 1 Drop of the ROP Study Drug | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | 1 Drop of the ROP Study Drug | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/43
Other Adverse Events (participants affected / at risk) | 0/40 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes